CLINICAL TRIAL: NCT00985647
Title: Pharmacokinetics of Plasma Lamivudine (3TC), and Its Active Intracellular Anabolite 3TC-Triphosphate Over a 24 Hour Dosing Interval Following Administration of 3TC 300 mg and 150 mg Once Daily to HIV-Negative Healthy Volunteers
Brief Title: Pharmacokinetics of Lamivudine at Two Different Doses
Acronym: ENCORE2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Marta Boffito, HIV/GUM Research Unit
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCHECR-ENCORE2
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections
Keywords: HIV; HAART; ART; Pharmacokinetic; Healthy volunteers; 3TC; Lamivudine
MeSH Terms: conditions — HIV Infections | interventions — Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3TC 300mg/150mg (Active Comparator): Group 1: Participants will be administered 3TC 300 mg once daily orally for 10 days. A 10 day wash-out period will follow (days 11-20). From day 21, participants will be administered 3TC 150 mg once daily for 10 days
  Interventions: Drug: Lamivudine (3TC)
- 3TC 150mg/300mg (Active Comparator): Group 2: Participants will be administered 3TC 150 mg once daily orally for 10 days. A 10 day wash-out period will follow (days 11-20). From day 21, participants will be administered 3TC 300 mg once daily for 10 days
  Interventions: Drug: Lamivudine (3TC)

INTERVENTIONS:
Drug: Lamivudine (3TC) — 3TC 300mg/150mg participants will receive 3TC 300 mg (2 x 150 mg tablet) once daily for 10 days, washout for 10 days and then 3TC 150 mg (1 x 150 mg tablet) once daily for 10 days.
  3TC 150mg/300mg participants will receive 3TC 150 mg (1 x 150 mg tablet) once daily for 10 days, washout for 10 days and then 3TC 300 mg (2 x 150 mg tablet) once daily for 10 days.
  Other Names: Epivir

SUMMARY:
The purpose of the study is to measure the pharmacokinetics (how a drug is absorbed, distributed and eliminated from the body) of lamivudine (3TC) and its active component after 3TC is given at two different doses, 300mg and 150mg once daily.

DETAILED DESCRIPTION:
Lamivudine (3TC) has been approved by regulatory authorities for the treatment of HIV infection and the current licensed dose is 300 mg once daily. Clinical and pharmacokinetic (how a drug is absorbed, distributed and eliminated from your body) data suggest that the licensing dose could be reduced without compromising effectiveness. Lower drug doses could reduce the side-effects from the medication and would make 3TC more affordable.

This study will compare the pharmacokinetics, safety and tolerability of two different doses of 3TC in healthy volunteers. The study will take place at Chelsea and Westminster Hospital. Twenty four healthy HIV negative volunteers will be randomly allocated into two groups. Volunteers in Group 1 will start 300mg 3TC once daily for 10 days, followed by 10 days of not taking any 3TC (wash-out period). When the wash-out period ends, they will re-start 3TC at a dose of 150mg once daily for 10 days. Group 2 is similar except that they will start 150mg 3TC at the beginning of the study and 300mg 3TC after the wash-out period. Blood samples will be taken over a 24-hour period at the end of each dosing phase to measure the levels of 3TC in the blood and inside blood cells. Safety and tolerability of 3TC will be assessed by questions, physical examination and laboratory parameters. These will be performed at regular intervals during the treatment phases.

Healthy participants as determined by their medical history and physical examination will be eligible to participate in the study. HIV-positive participants will not be recruited because it is not yet clear if an experimentally reduced dose of 3TC will successfully treat HIV-infection. There is no reason to presume that there is any meaningful difference in the metabolic processing of 3TC between HIV-infected and HIV-uninfected people.

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
2. Male or non-pregnant, non-lactating females
3. Between 18 to 65 years, inclusive
4. Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive
5. Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 1 month after the study.

Exclusion Criteria:

1. Any significant acute or chronic medical illness
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
3. Positive blood screen for hepatitis B core and/or C antibodies and/or hepatitis B surface antigen
4. Positive blood screen for HIV-1 and/or 2 antibodies
5. Current or recent (within 3 months) gastrointestinal disease
6. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study
7. Exposure to any investigational drug or placebo within 3 months of first dose of study drug
8. Use of any other drugs, including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs
9. Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 30 days after the end of the treatment period
10. Previous allergy to any of the constituents of the pharmaceuticals administered in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of 3TC and intracellular concentrations of its active anabolite 3TC-TP as measured by the Area Under the Curve (AUC 0-24h). | Measured over 24 hours at the end of each 10-day dosing period.
  Concentrations will be compared after the administration of 3TC 300 mg and 150 mg once daily.

SECONDARY OUTCOMES:
Safety and tolerability of 3TC following the administration of 3TC 300 mg and 150 mg once daily | Assessed at regular intervals throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, MD PhD, Principal Investigator — Chelsea and Westminster Hospital
Locations (1):
- St Stephen's Centre, Chelsea and Westminster Hospital, London, United Kingdom